CLINICAL TRIAL: NCT05643729
Title: A Phase I/II Randomized, Double Blinded, Placebo Trial to Evaluate the Safety and Potential Efficacy of Intravenous Infusion (IV) of ZofinTM for the Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Zofin to Treat Chronic Obstructive Pulmonary Disease (COPD)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is on hold
Sponsor: ZEO ScientifiX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27198
Record Dates: First submitted 2022-11-01; First posted 2022-12-09 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-10

CONDITIONS: COPD
Keywords: Zofin; Human Amniotic Fluid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a phase I/II randomized, double blinded and placebo control. The ratio between groups is 1:1 for total 20 subjects. Each subject will be randomized to receive either treatment or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be double blinded such that neither the patients nor the researchers will know who is getting a placebo and who is getting the treatment. Only product manufacturing staff will be un-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Zofin (Experimental): Group 1 Treatment Arm (10 subjects): Zofin + Standard of care (SOC) Ten subjects will receive 1 mL of Zofin on Day 0, Day 4, and Day 8, containing 1-5 x 10^11 particles/ml. The Zofin dose will be diluted in 100 mL of sterile saline at subject's bedside. In addition to Zofin all subjects in this trial will receive SOC throughout the study period.
  Interventions: Drug: Zofin
- Group 2: Placebo (Placebo Comparator): Group 2 Control Arm (10 subjects): Placebo + SOC Ten subjects will receive placebo on Day 0, Day 4, and Day 8, containing 101 mL of sterile saline at subject's bedside. In addition to placebo all subjects in this trial will receive SOC throughout the study period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zofin — Intravenous Infusion (IV) of Zofin
  Arms: Group 1: Zofin
Other: Placebo — Intravenous Infusion of sterile saline
  Arms: Group 2: Placebo

SUMMARY:
A Phase I/II Randomized, Double Blinded, Placebo Trial to Evaluate the Safety and Potential Efficacy of Intravenous Infusion (IV) of Zofin for the Treatment of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Total of 20 adult patients will be chosen from population of adults between the age of 40 to 80 diagnosed with COPD to be randomized to 1 of 2 treatment arms including IV infusion of Zofin or IV infusion on sterile saline.

The subjects will be followed for 12 months to demonstrate safety and efficacy of Zofin.

ELIGIBILITY:
Inclusion Criteria:

* Subject who can understand and are able to provide informed consent.
* Subject with moderate to severe COPD with normal cardiac, liver and renal function
* Subject must have a post-bronchodilator FEV1/FVC ratio of less than 0.7
* Subject must have a post-bronchodilator FEV1 percent predicted value <50%
* Subject must have a RV/TLC ratio of > 40%
* Subject must be either a non-smoker or an ex-smoker, with a cigarette smoking history of ≥ 10 packs per year.
* Subject must have abstained from nicotine products for at least six months prior to enrollment in the study.
* Subject must be available for all specified assessments at the study site through the completion of the study.
* Subject must have oxyhemoglobin saturation on room air at rest equal or greater than 88% without oxygen
* Subject must be reasonably able to return for multiple follow-up visits.
* Adequate venous access
* For Women of Child-Bearing Potential (WOCBP) only, willingness to use FDA-recommended birth control until 6 months post treatment.
* Any male subject must agree to use contraceptives and not donate sperm during the study.

Exclusion Criteria:

* Subject with clinically significant illness with manifestations of significant organ dysfunction which in the judgment of the PI or co-investigator would render the study subject unlikely to tolerate the infusion or complete the study

  * Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening which will be within 72 hours of the IP infusion.
  * Subject has been diagnosed with a pulmonary disease other than COPD (e.g. asthma, pulmonary, fibrosis, sarcoidosis, pulmonary hypertension, bronchiolitis, interstitial lung disease)
  * Subject has been diagnosed with α1-Antitrypsin deficiency
  * Subject has a body mass index greater than 42 kg/m2
  * Subject has or had an active infection requiring systemic antibiotics within 12 weeks on enrollment in the study
  * Subject has or had exacerbation of COPD requiring hospitalization within 12 weeks of enrollment in the study.
  * Subject has initiated pulmonary rehabilitation within 12 weeks of enrollment in the study
  * Subject uses or used prednisone (or equivalent dose of another corticosteroid) within 12 weeks of enrollment in the study
  * Subject has evidence or history of malignancy
  * Subject has evidence or history of autoimmune disorders independent of COPD
  * Subject is pregnant or breast-feeding
  * Subject with pulmonary lobectomy or lung volume reduction surgery or lung transplantation. Subject with clinically significant bronchiectasis.
  * Subject received an experimental therapy (drug or biologic) for any indication within 12 months of the study enrollment.
  * Subject is unable to complete all the testing required for the study
  * Subject who is on immunosuppressive medications.
  * Subject who is unwilling to stop taking prescription or over the counter pain medication for 7 days prior to any visit.
  * Subject with a history of bleeding disorders, anticoagulation therapy that cannot be stopped as prior to infusion.
  * Active listing (or expected future listing) for transplant of any organ.
  * Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
  * History of drug abuse (illegal "street" drugs) except noninhalation use of marijuana (If it is legal use in states where patient resides), or prescription medications not being used appropriately for a pre-existing medical condition or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs withinthe past 24 months. Use of inhalation marijuana will be an exclusion criterion.
  * Subject with untreated HIV infection. However, patients can be enrolled if they have been treated for HIV and test negative for HIV viral load but still test positive for antibodies.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Zofin | first 30 days
  To demonstrate the safety of Zofin administered intravenously in subjects with COPD by measuring incidence of any of the following treatment-emergent serious adverse events (TE-SAEs) within the first 30 days of infusion:
  * Life-threatening event (e.g., stroke or non-fatal pulmonary embolism).
  * Event requiring inpatient hospitalization or prolongation of existing hospitalization (e.g., for worsening dyspnea).
  * Event resulting in persistent or significant disability/incapacity.
  * Event resulting in death. Frequency and severity of any adverse events from Day 0 (day of treatment) up to 12 months of treatment will similarly be observed.
Safety of Zofin | day 0 to 12 months
  To monitor the frequency and severity of adverse events

SECONDARY OUTCOMES:
FVC | Screen, day 4, day 8, 4 months, 8 months and 12 months
  FVC from resting PFT
FEV1 | Screen, day 4, day 8, 4 months, 8 months and 12 months
  FEV1 from resting PFT
FEV1 to FVC ratio | Screen, day 4, day 8, 4 months, 8 months and 12 months
  FEV1 to FVC ratio on resting pulmonary function test
FEF25-75 | Screen, day 4, day 8, 4 months, 8 months and 12 months
  FEF25-75 on resting pulmonary function test
Lung Volume Changes | Screen, day 4, day 8, 4 months, 8 months and 12 months
  Change in lung volumes (in body plethysmograph), including SGAW (specific airway conductance) and RV (to calculate gas trapping)
DLCO | Screen, day 4, day 8, 4 months, 8 months and 12 months
  Change in single breath diffusing capacity of lung for carbon monoxide (DLCO)
HU of CT Scan | Screen and 12 months
  Change in the average of Hounsfield Unit (HU) - a relative quantitative measurement of radio density in CT images.
% air in lung on CT Scan | Screen and 12 months
  Change in the percentage of air in the lung
CPET | Screen, 4 months, and 12 months
  Cardiopulmonary Exercise Testing (CPET) with peak VO2 and measures of dynamic hyperinflation
Peak VO2 | Screen, 4 months, and 12 months
  Cardiopulmonary Exercise Testing (CPET) with peak VO2
Dynamic Hyperinflation | Screen, 4 months, and 12 months
  Cardiopulmonary Exercise Testing (CPET) with measures of dynamic hyperinflation
Pulmonary Exacerbation | Screening through 12 months
  Incidence of investigator-defined pulmonary exacerbation: decrease in exacerbation-related hospitalization
TNF-α | Day 0, Day14, 4 months, 8 months, and 12 months
  Change in serum inflammatory markers: TNF-α
CRP | Day 0, Day14, 4 months, 8 months, and 12 months
  Change in serum inflammatory markers: CRP
IL-1 | Day 0, Day14, 4 months, 8 months, and 12 months
  Change in serum inflammatory markers: IL-1
D-Dimer | Day 0, Day14, 4 months, 8 months, and 12 months
  Change in serum inflammatory markers: D-dimer
Fibrinogen | Day 0, Day14, 4 months, 8 months, and 12 months
  Change in serum inflammatory markers: Fibrinogen
SF-36 ot SGRQ | Screen, 14 days, 1.5 months, 4 months, 8 months, and 12 months
  Change in SF-36 questionnaire or St. George's Respiratory Questionnaire (SGRQ)
CAT Assessment | Screen, 14 days, 1.5 months, 4 months, 8 months, and 12 months
  Change in quality of life (QOL) assessments via COPD Assessment Test (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Phrsai, Study Director — Proxima
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No